CLINICAL TRIAL: NCT00377845
Title: Cervix Cytological Screening - Comparison of Tampon Self-Test and the Routine Smear.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Else Toft Würtz, Student
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: TP06-2351
Record Dates: First submitted 2006-09-18; First posted 2006-09-19 (Estimated); Last update posted 2008-03-27 (Estimated); Status verified 2008-03

CONDITIONS: Uterine Cervical Dysplasia; Uterine Cervical Neoplasms
Keywords: self test; PAP smear; tampon test; cervical dysplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Regular Tampax used in 3 hours

SUMMARY:
The purpose of this study is to compare suitability, specificity and sensitivity of the routine smear and the tampon self-test women perform at home.

Study hypothesis: The tampon self-test correspond to the routine cervical smear.

ELIGIBILITY:
Inclusion Criteria:

1. Women with cervical dysplasia been referred to conisation or
2. Women invited to cervical screening program

Exclusion Criteria:

1. Women not performing the tampon self-test before conisation or
2. Women not performing the tampon self-test af least 1 month after receiving the tampon

Min Age: 23 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-09; Primary Completion 2007-12 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the tampon self-test

SECONDARY OUTCOMES:
The womens socio-demographic relations according to accept the tampon self-test

CONTACTS AND LOCATIONS:
Overall Officials: Hans Svanholm, consultant, Study Director — Randers Hospital, Pathological Institute
Locations (1):
- Region Hospital Randers, Randers, Denmark